CLINICAL TRIAL: NCT05894044
Title: Effects of Different Modalities of Medium and Low Frequency Electrical Stimulation in the Generation of Evoked Torque, Sensory Discomfort, Muscle Fatigue and Inheritance Peripheral Oxygen Supply in the Triceps Surae Muscle.
Brief Title: Effects of Kilohertz-frequency and Low-frequency Current on Triceps Surae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 67915523.1.0000.8093
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Electrical stimulation; Burst; M-wave; H-reflex; Pulsed current; Russian current; Aussie Current

STUDY DESIGN:
Intervention Model Description: This is a crossover, experimental, randomized, double-blind trial composed of apparently healthy participants.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Russian current 10% (Experimental): Subjects will receive a interventions (Russian Current at 10% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Russian current 10%
- Aussie current 10% (Experimental): Subjects will receive a interventions (Aussie Current at 10% duty cycle). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Aussie current 10%
- Pulsed current 500 µs phase (Experimental): Subjects will receive a interventions (Pulsed current with 50 Hz, 500 µs phase). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Pulsed current 500 µs phase
- Pulsed current 200 µs phase (Experimental): Subjects will receive a interventions (Pulsed current with 50 Hz, 200 µs phase). Evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction will be evaluated.
  Interventions: Other: Pulsed current 200 µs phase

INTERVENTIONS:
Other: Russian current 10% — Russian current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts
  Other Names: Russian current with 2500 Hz, modulated in bursts of 50 Hz, 200 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts
  Arms: Russian current 10%
Other: Aussie current 10% — Aussie current with 1000 Hz, modulated in bursts of 50 Hz, 500 µs and 10% duty cycle - 2 ms bursts and 18 ms interbusrts
  Arms: Aussie current 10%
Other: Pulsed current 500 µs phase — Pulsed current, modulated in 50 Hz, 500 µs
  Arms: Pulsed current 500 µs phase
Other: Pulsed current 200 µs phase — Pulsed current, modulated in 50 Hz, 200 µs
  Arms: Pulsed current 200 µs phase

SUMMARY:
Neuromuscular electrical Stimulation (NMES) can minimize muscle atrophy and complications related to muscle disuse and help improve neuromuscular performance. Medium and low-frequency currents have been assessed regarding the generation of evoked torque, sensory discomfort, muscle fatigue, and peripheral oxygen extraction. In addition, metabolic stress is also linked to muscle strength gain, an important aspect to be evaluated in addition to NMES physical parameters. Thus, the aim of this study is to compare the effects of different NMES protocols applied to the triceps surae muscle for evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction in healthy individuals. This is a crossover, experimental, randomized, double-blind trial composed of apparently healthy participants. All NMES protocols will be tested on the same individual with randomization of the sequence of intervention protocols. There will be a total of 5 encounters with seven days between them. Session 1 will evaluate the anthropometric measures, the maximum intensity for each intervention protocol, and the sequence of intervention protocols for each individual will be randomized. Sessions 2, 3, 4, and 5 will be composed equally with the assessment of the maximum voluntary and evoked joint torque of the triceps surae muscle through the isokinetic dynamometer, evaluation of muscle fatigue through the H-reflex, M-wave, fatigue index, time-torque-integral, and recruitment curve, evaluation of peripheral oxygen extraction through NIRS (Near Infrared Spectroscopy), electromyographic signals to assessed the RMS (root mean square) and the median frequency, evaluation of the level of sensory discomfort through the Visual Analog Pain Scale and finally by the NMES protocol. The EENM protocols will be as follows: CR10% (Russian Current at 2500 Hz, modulated in 50 Hz bursts, 200 µs and 10% duty cycle - 2 ms of 18 ms bursts and interbusrts), CA10% (Aussie Current with 1000 Hz, modulated in 50 Hz bursts, 500 µs and 10% duty cycle - 2 ms of 18 ms bursts and interbusrts), CP500 (pulsed current with 50 Hz, 500 µs phase) and CP200 (Pulsed current with 50 Hz, 200 µs phase). all protocols will be performed on the triceps surae muscle.

DETAILED DESCRIPTION:
This is a crossover, experimental, randomized, double-blind trial composed of apparently healthy participants. The objective is to compare the effects of different NMES protocols applied to the triceps surae muscle for evoked torque, muscle fatigue, sensory discomfort, and peripheral oxygen extraction. The effects of the types of neuromuscular electrical stimulation (NMES) protocols on the aforementioned outcomes will be evaluated in the same participant by randomizing the sequences of interventions for each visit in the laboratory. The study is considered double-blind, as individuals will not know the sequence of the protocols applied. The evaluator will also not know which protocol will be used at the time of the intervention. It will consist of a total of 5 sessions with seven days between them. In the first session, anthropometry, the maximum intensity level for each electrical stimulation protocol as well as the protocol sequence for each individual will be evaluated. From the second to the fifth session, the following will be considered: voluntary and evoked maximum joint torque of the triceps surae muscle, muscle fatigue through the evaluation of the H-reflex, M-wave, fatigue index, torque-time-integral and recruitment curve, peripheral oxygen extraction, electromyographic signals through RMS (root mean square) and median frequency, and level of sensory discomfort with the Visual Analog Scale (VAS). From the second to the fifth session will be composed by the following evaluation sequence: warm-up with six submaximal contractions with 6 seconds of duration and 10 seconds of rest between them; then the assessment of muscle fatigue; then two maximal isometric contractions, then two maximal evoked contractions; fatigue protocol at 20% of the maximum isometric contraction (this fatigue protocol will use the NMES sequence randomized in the first session; after the fatigue protocol, two maximum evoked contractions will be performed again; then two maximal isometric contractions and at the end, the muscle fatigue evaluation will be performed again. The NMES protocols will be CR10% (Russian Current at 2500 Hz, modulated in 50 Hz bursts, 200 µs and 10% duty cycle - 2 ms of 18 ms bursts and interbusrts), CA10% (Aussie Current with 1000 Hz, modulated in 50 Hz bursts, 500 µs and 10% duty cycle - 2 ms of 18 ms bursts and interbusrts), CP500 (pulsed current with 50 Hz, 500 µs phase) and CP200 (Pulsed current with 50 Hz, 200 µs phase). All protocols will be performed on the triceps surae muscle.

ELIGIBILITY:
Inclusion Criteria:

* Female and male, aged between 18-40 years;
* Be classified as physically active according to the International Physical Activity Questionnaire (IPAQ);
* The practice of just recreational physical activity;
* Achieve a minimum torque of 20% of the MVIC during the NMES;
* Be at least three months without strength training;

Exclusion Criteria:

* Present musculoskeletal dysfunction that may interfere with the tests, present intolerance to NMES in the triceps surae muscle;
* Use analgesics, antidepressants, tranquilizers, or other centrally acting agents;
* Present cardiovascular or peripheral vascular problems, chronic diseases, neurological or muscle disorders that may impair the complete execution of the study design by the volunteer;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Submaximal voluntary isometric contraction of the triceps surae | 2 minutes
  Expressed in muscle strength, assessed using an isokinetic dynamometer
Maximum voluntary isometric contraction of the triceps surae | 5 minutes
  Expressed in muscle strength, assessed using an isokinetic dynamometer
Maximum evoked torque | 5 minutes
  Expressed by the description of muscle strength generated by electrical stimulation assessed by the isokinetic dynamometer
Torque evoked during the fatigue protocol | 15 minutes
  Expressed by the description of muscle strength generated by electrical stimulation assessed by the isokinetic dynamometer
Muscle fatigue assessment before the muscle fatigue protocol | 10 minutes
  Expressed by mechanical properties of plantar flexors and central activation relationship using the contraction interpolation technique
Assessment of muscle fatigue during the muscle fatigue protocol | 20 minutes
  Expressed by the muscle fatigue index through the decline in torque evoked from the beginning to the end of the protocol
Muscle fatigue assessment during the muscle fatigue protocol | 20 minutes
  Expressed by the decline in torque-time-integral from the beginning to the end of the protocol

SECONDARY OUTCOMES:
Sensory discomfort during maximum evoked torques | 10 seconds
  Measured through the Visual Analog Scale (1 - 10 cm) where 0 represents no discomfort and 10 represents greater discomfort
Sensory discomfort during fatigue protocol | 10 seconds
  Measured through the Visual Analog Scale (1 - 10 cm) where 0 represents no discomfort and 10 represents greater discomfort
Electromyographic signals | 40 minutes
  Expressed by the raw values of RMS and Median Frequency within a range of 500 ms throughout the entire session
Peripheral oxygen extraction | 40 minutes
  Expressed by peripheral oxygen consumption assessed by near-infrared spectroscopy from the beginning to the end of the sessions

CONTACTS AND LOCATIONS:
Overall Officials: João LQ Durigan, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Faculty of Ceilandia UnB, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No
The authors consider sharing the data depending on the situation.

REFERENCES:
- [Background] Baldi JC, Jackson RD, Moraille R, Mysiw WJ. Muscle atrophy is prevented in patients with acute spinal cord injury using functional electrical stimulation. Spinal Cord. 1998 Jul;36(7):463-9. doi: 10.1038/sj.sc.3100679. PMID 9670381
- [Background] Ward AR, Lucas-Toumbourou S, McCarthy B. A comparison of the analgesic efficacy of medium-frequency alternating current and TENS. Physiotherapy. 2009 Dec;95(4):280-8. doi: 10.1016/j.physio.2009.06.005. Epub 2009 Sep 2. PMID 19892092
- [Background] Aldayel A, Jubeau M, McGuigan M, Nosaka K. Comparison between alternating and pulsed current electrical muscle stimulation for muscle and systemic acute responses. J Appl Physiol (1985). 2010 Sep;109(3):735-44. doi: 10.1152/japplphysiol.00189.2010. Epub 2010 Jul 1. PMID 20595542
- [Background] Arpin DJ, Forrest G, Harkema SJ, Rejc E. Submaximal Marker for Investigating Peak Muscle Torque Using Neuromuscular Electrical Stimulation after Paralysis. J Neurotrauma. 2019 Mar 19;36(6):930-936. doi: 10.1089/neu.2018.5848. Epub 2018 Nov 16. PMID 30226407
- [Background] Martin A, Grospretre S, Vilmen C, Guye M, Mattei JP, LE Fur Y, Bendahan D, Gondin J. The Etiology of Muscle Fatigue Differs between Two Electrical Stimulation Protocols. Med Sci Sports Exerc. 2016 Aug;48(8):1474-84. doi: 10.1249/MSS.0000000000000930. PMID 27031743
- [Background] Neyroud D, Dodd D, Gondin J, Maffiuletti NA, Kayser B, Place N. Wide-pulse-high-frequency neuromuscular stimulation of triceps surae induces greater muscle fatigue compared with conventional stimulation. J Appl Physiol (1985). 2014 May 15;116(10):1281-9. doi: 10.1152/japplphysiol.01015.2013. Epub 2014 Mar 27. PMID 24674861
- [Background] Pinto Damo NL, Modesto KA, Neto IVS, Bottaro M, Babault N, Durigan JLQ. Effects of different electrical stimulation currents and phase durations on submaximal and maximum torque, efficiency, and discomfort: a randomized crossover trial. Braz J Phys Ther. 2021 Sep-Oct;25(5):593-600. doi: 10.1016/j.bjpt.2021.03.001. Epub 2021 Mar 26. PMID 33840592
- [Background] da Silva VZ, Durigan JL, Arena R, de Noronha M, Gurney B, Cipriano G Jr. Current evidence demonstrates similar effects of kilohertz-frequency and low-frequency current on quadriceps evoked torque and discomfort in healthy individuals: a systematic review with meta-analysis. Physiother Theory Pract. 2015;31(8):533-9. doi: 10.3109/09593985.2015.1064191. Epub 2015 Oct 14. PMID 26467544
- [Background] Bellew JW, Cayot T, Brown K, Blair C, Dishion T, Ortman B, Reel A. Changes in microvascular oxygenation and total hemoglobin concentration of the vastus lateralis during neuromuscular electrical stimulation (NMES). Physiother Theory Pract. 2021 Aug;37(8):926-934. doi: 10.1080/09593985.2019.1652945. Epub 2019 Aug 12. PMID 31402741